CLINICAL TRIAL: NCT02197156
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Active Comparator Study of Hydrocodone Bitartrate Extended Release (HC-ER) in Adults Following Bunionectomy Surgery
Brief Title: A Multicenter Active Comparator Study of HC-ER in Adults Following Bunionectomy Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ELN154088-201
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2014-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 10 mg HC-ER (Experimental): Hydrocodone bitartrate extended release (HC-ER) 10 mg
  Interventions: Drug: 10 mg HC-ER
- 20 mg HC-ER (Experimental): Hydrocodone bitartrate extended release (HC-ER) 20 mg
  Interventions: Drug: 20 mg HC-ER
- 30 mg HC-ER (Experimental): Hydrocodone bitartrate extended release (HC-ER) 30 mg
  Interventions: Drug: 30 mg HC-ER
- 40 mg HC-ER (Experimental): Hydrocodone bitartrate extended release (HC-ER) 40 mg
  Interventions: Drug: 40 mg HC-ER
- 10 mg HC / 325 mg APAP (Active Comparator): 10 mg Hydrocodone (HC) / 325 mg acetaminophen (APAP)
  Interventions: Drug: 10 mg HC / 325 mg APAP
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: 10 mg HC-ER — Single dose
  Other Names: ELN154088; Hydrocodone bitartrate extended release (HC-ER); Zohydro Extended Release (ER)
  Arms: 10 mg HC-ER
Drug: 20 mg HC-ER — Single dose
  Other Names: ELN154088; Hydrocodone bitartrate extended release (HC-ER) 10 mg; Zohydro Extended Release (ER)
  Arms: 20 mg HC-ER
Drug: 30 mg HC-ER — Single dose
  Other Names: ELN154088; Hydrocodone bitartrate extended release (HC-ER) 30 mg; Zohydro Extended Release (ER)
  Arms: 30 mg HC-ER
Drug: 40 mg HC-ER — Single dose
  Other Names: ELN154088; Hydrocodone bitartrate extended release (HC-ER) 40 mg; Zohydro Extended Release (ER)
  Arms: 40 mg HC-ER
Drug: 10 mg HC / 325 mg APAP — Single dose
  Other Names: 10 mg Hydrocodone (HC) / 325 mg acetaminophen (APAP)
  Arms: 10 mg HC / 325 mg APAP
Drug: Matching Placebo — Single dose
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to establish a dose-response relationship among several capsule strengths of Hydrocodone Bitartrate Extended Release (HC-ER) and to compare the efficacy to placebo following bunionectomy surgery

DETAILED DESCRIPTION:
Sum of Pain Intensity Differences (SPID) for the Primary pain measurement: VASPI (Visual Analog Scale of Pain Intensity) from time 0 to 12 hrs; Safety evaluations assessed: laboratory evaluations, physical examinations, vital signs/pulse oximetry and electrocardiography

ELIGIBILITY:
Inclusion Criteria:

* Subject was able to read and voluntarily sign the Institutional Review Board (IRB) approved, written informed consent document and given the opportunity to ask questions regarding the study prior to the performance of any study- specific procedures.
* Subject required primary unilateral first metatarsal bunionectomy surgery with or without hammertoe repair with no other collateral procedures allowed
* Subject was male or female at least 18 years of age.
* Subject weighed > or = 100 lbs (pounds).
* Subject was willing and able to comply with the protocol and able to score their pain intensity.
* Subject was in good health as determined by the investigator on the basis of medical history, physical examination, Electrocardiogram (ECG) and screening laboratory results.
* Subject had not developed a condition or complications as result of the bunionectomy procedure that would preclude their participation in the study.
* Subject was willing and able to remain at the recovery day care center for the entire 24-hour Treatment period.

Exclusion Criteria:

* Subject was pregnant or lactating.
* Subject had been on an investigational drug within 30 days prior to the initiation of study drug.
* Subject had donated blood or blood components within one month prior to study (Check-in).
* Subject had a know allergy or hypersensitivity to opioids, acetaminophen, and/or ketorolac.
* Subject had a known history of substance or alcohol abuse within 2 years prior to Screening.
* Subject tested positive to drug screens (cocaine, marijuana, opioids, benzodiazepines, and barbiturates) that could not be justified by prescription use.
* Subject had a condition that would contraindicate the use of opioid analgesia (e.g., pulmonary disease or paralytic ileus).
* Subject had received a selective serotonin reuptake inhibitor (SSRI), monoamine oxidase inhibitor (MAOI) carbamazepine, quinidine, and/or tricyclic antidepressants (TCA) compounds within 1-month prior to Check-in.
* Subject had received opioids, tranquilizers, sedatives, or hypnotics within 48 hours prior to Check-in.
* Subject had received corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or other analgesics within 24 hours prior to Check-in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2002-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
The Sum of Pain Intensity Differences (SPID) for the Visual Analog Scale Pain Intensity (VASPI) | 0-12 hours